CLINICAL TRIAL: NCT04114227
Title: Acceptance and Commitment Therapy vs. Supportive Psychotherapy With Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, C. Virginia O'Hayer, Principal Investigator, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1905007203
Record Dates: First submitted 2019-09-23; First posted 2019-10-03 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Active Comparator): Participants will learn new ways to manage uncomfortable experiences and feelings and to engage in positive behaviors.
  Interventions: Behavioral: Acceptance and Commitment Therapy adapted for Cystic Fibrosis (ACT with CF)
- Supportive Psychotherapy (Active Comparator): Participants will talk about their experiences to date.
  Interventions: Behavioral: Supportive Psychotherapy (Treatment as Usual Control)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy adapted for Cystic Fibrosis (ACT with CF) — Subjects learn new ways to manage uncomfortable experiences and feelings and to engage in positive behaviors
  Arms: Acceptance and Commitment Therapy
Behavioral: Supportive Psychotherapy (Treatment as Usual Control) — Subjects talk about their experiences to date in a cohort of adult Cystic Fibrosis patients.
  Arms: Supportive Psychotherapy

SUMMARY:
The objective of the study is to assess the utility of "Acceptance and Commitment Therapy" (ACT) in which subjects learn new ways to manage uncomfortable experiences and feelings and to engage in positive behaviors, over "Supportive Psychotherapy" in which subjects talk about their experiences to date in a cohort of adult Cystic Fibrosis patients. The hypothesis is that six telehealth/webcam sessions of ACT will lead to an improvement in medication and visit compliance, as well as an overall improved sense of well-being and coping skills, particularly as compared with 6 telehealth/webcam sessions of supportive psychotherapy.

DETAILED DESCRIPTION:
Patients will be consented in the adult cystic fibrosis clinic at Drexel University, Children's Hospital of Philadelphia, University of Pennsylvania Medical Center, St. Christopher's Hospital for Children, Duke University Medical Center, Augusta University and the University of Pittsburgh. For Philadelphia sites (CHOP, Drexel, UPenn, St. Chris), Chelsi Nurse will consent patients to treatment. If at remote sites (Duke Univ Med Center, Augusta Univ, U Pittsburgh) by our local site appointed representatives will consent patients to the study. All CF patients will be approached to assess interest.

If patients are willing to be in the study, they will be given a packet of screening questionnaires (addendum #1). These questionnaires will ask patients: 1) how often participants experience different thoughts and feelings, including some related to having cystic fibrosis; 2) how often participants take their cystic fibrosis medications; 3) their coping style, including how long participants persist in thinking about something that has happened to them; The subject will complete each questionnaire again after 6 appointments (i.e., about 6 weeks later), and again about 3-months after their sixth appointment.

Finally, the investigators hope to learn whether these therapies affect how often subjects take their cystic fibrosis medications, and how this affects their health and wellbeing.

To study this, the investigators will review the number of appointments that are missed six months before enrolling in the program, and six months after completing therapy.The investigators will also review their pulmonary function tests, whether subjects go to the hospital or see their doctor for any extra visits, and the presence of any ongoing symptoms of depression or anxiety. All data will be taken from Allscripts, the Drexel outpatient medical chart. Data will be taken only from the departments of the pi and co-pi's. At UPenn, the social worker at the site will input data into Drexel Redcap through a link sent to them.

Participants will complete 6 sessions of our ACT with CF manualized intervention. Participants will be asked to complete a series of brief questionnaires at the time of consent. If desired, they can take these homes to complete and mail back.

These questionnaires will ask participants about: 1) how often they experience different thoughts and feelings, including some related to having cystic fibrosis; 2) how often they take their cystic fibrosis medications; 3) their coping style, including how long they persist in thinking about something that has happened to them.

Participants will complete each questionnaire again after 6 appointments (i.e., about 6 weeks later), and again about 3-months after their sixth appointment.

These questionnaires take about 45 minutes to complete. Participants will also be asked to complete 6 'Zoom' therapy sessions (using a webcam in their own home or on their own tablet/smartphone and HIPAA-compliant Zoom webcam service) of either "Acceptance and Commitment Therapy", in which participants will learn new ways to manage uncomfortable experiences and feelings (e.g., depression, anxiety) and to engage in positive behaviors, or to "Supportive Psychotherapy", in which participants will talk about their experiences to date. The type of therapy that participants get will be chosen by chance, like flipping a coin. Neither subject nor the study doctor will choose what treatment the participant will get. Participants will have an equal chance of being given each therapy. Audio and video recordings will be taken during each 'Zoom' therapy session. Recordings will be kept on password encrypted USB drives and stored in a locked office only accessible to the principal investigator and adherence coder. Finally, the investigators hope to learn whether these therapies affect how often participants take their cystic fibrosis medications, and how this affects their health and wellbeing. To study this, the investigators will review information from medical charts such as the number of appointments that kept, the number of appointments missed, pulmonary function tests, number of hospital or doctor visits, and the presence of any symptoms of depression or anxiety.

Measures administered are as follows:

Page 1-2: Demographics Page 3-6: CFMHWQ: CF Mental Health and Wellness Self-Report Measure. Page 7-8: BDI-II: Beck Depression Inventory-II. Page 9: BAI: The Beck Anxiety Index. Pearson. Page 10-13: CFQ-R: Cystic Fibrosis Questionnaire-Revised. Page 14: Medical Coping Modes Questionnaire. Page 15: CFS: Coping Flexibility Scale. Page 16: My CF Treatments: Treatment Adherence Questionnaire-CF. Page 17-18: ACT Demographics Page 19: CFQ13: Cognitive Fusion Questionnaire. Page 20: Short Grit Scale Page 21: AAQ-II: Acceptance and Action Questionnaire. Page 22-23: Styles of Coping Word-Pairs.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and above.
* Able to read/understand English.
* Diagnosis of cystic fibrosis.
* PHQ-9 score > 4 or GAD-7 score > 4.

Exclusion Criteria:

* History of suicidal attempts or acute suicidal ideation on clinical assessment.
* Presence of psychotic disorder or symptoms.
* Pregnant women.
* Presence of psychiatric disorders that interfere with the participation of the study, judged by the study or treating clinician. Presence of other medical conditions that interfere with participation in the study, judged by the study or treating clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Change at baseline (study entry point, before any sessions have been delivered), after 6 weeks of treatment, 3 months after the end of 6 sessions of treatment.
  This scale is a self-report measure of anxiety.
Beck Depression Inventory-II (BDI-II) | Change at baseline (study entry point, before any sessions have been delivered), after 6 weeks of treatment, 3 months after the end of 6 sessions of treatment.
  Widely used indicator of the severity of depression.
Cognitive Fusion Questionnaire (CFQ13) | Beginning of study, after 6 weeks, after 3 months.
  Change in cognitive fusion (rigid attachment to one's thoughts as Truth) measures.
Acceptance and Action Questionnaire (AAQ-II) | Beginning of study, after 6 weeks, after 3 months.
  Change in acceptance measures.

SECONDARY OUTCOMES:
FEV1/ FVC ratio | 3 months before study, 3 months after study.
  Change in FEV1/FVC ratio.
The Treatment Adherence Questionnaire-CF | Beginning of study, after 6 weeks, after 3 months.
  Participant change in medication adherence.
The Cystic Fibrosis Questionnaire-Revised (CFQ-R) | Beginning of study, after 6 weeks, after 3 months.
  Change in CF-related quality of life

OTHER OUTCOMES:
Generalized Anxiety Disorder Questionnaire 7 (GAD-7) | Inclusion screening measure
  Rapid screening for the presence of a clinically significant anxiety disorder.
Patient Health Questionnaire 9 (PHQ-9) | Inclusion screening measure
  Use as a screening tool to assist the clinician in making the diagnosis of depression and to quantify depression symptoms and monitor severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Jefferson Center City Clinic for Behavioral Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith PJ, Drescher CF, Bruschwein H, Ingle K, Nurse C, O'Hayer CV. Psychological Flexibility, Coping Styles, and Mood Among Individuals With Cystic Fibrosis. Biopsychosoc Sci Med. 2025 May 1;87(4):271-279. doi: 10.1097/PSY.0000000000001387. Epub 2025 Mar 24. PMID 40167140
- [Derived] O'Hayer CV, Smith PJ, Drescher CF, Bruschwein H, Nurse CN, Kushner HM, Ingle K, Stephen MJ, Hoag JB. ACT with CF: A randomized trial of acceptance and commitment therapy vs supportive psychotherapy for adults with cystic fibrosis. Gen Hosp Psychiatry. 2024 Nov-Dec;91:212-222. doi: 10.1016/j.genhosppsych.2024.11.011. Epub 2024 Nov 26. PMID 39626332

DOCUMENTS (2):
  • Study Protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04114227/Prot_000.pdf
  • Informed Consent Form (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT04114227/ICF_001.pdf